CLINICAL TRIAL: NCT07309653
Title: Colour Matching, Stability, and Patient's Satisfaction in Maxillary Anterior Restorations Using Single-Shade Composite and Silicone-Guided Index: A 12-Month Clinical Evaluation
Brief Title: Colour Match, Stability, and Patient's Satisfaction of Single-Shade Composites in Anterior Teeth
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sawanya Prutthithaworn, Principal Investigator, Mahidol University
Other Study IDs: MU-DT/PY-IRB 2025/082.3010
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Tooth Injuries; Dental Restoration, Permanent
Keywords: Patient satisfaction; Color stability; Color matching; Single shade composter resins; Injection moulding technique; Flowable composite resins; Dental trauma
MeSH Terms: conditions — Tooth Injuries; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test: Restoring with an injectable single shade composite resin using an injectable moulding technique

SUMMARY:
The goal of this observational study is to evaluate the clinical performance of a single-shade composite resin, used with an injection moulding technique, in restoring maxillary incisors affected by traumatic dental injury in patients aged 6-15 years.

The main questions it aims to answer are:

* How well does a single composite resin colour match the natural tooth?
* How stable is the colour over a 6- and 12-month follow-up?
* How satisfied are the children and parents with the restoration?

ELIGIBILITY:
Inclusion Criteria:

* Children who exhibit cooperative dental behaviours (rating 3 and 4) according to Frankl's behaviour rating scale (Frankl et al. 1962)
* Presence of at least one maxillary anterior permanent tooth with one-third of crown structure loss from dental trauma
* The affected tooth must be vital or have undergone vital pulp therapy (e.g., pulpotomy with Calcium hydroxide, white-MTA, or Biodentine)

Exclusion Criteria:

* Known allergy to methacrylate-based materials
* Presence of parafunctional habits, such as bruxism
* Presence of rampant caries
* Presence of signs of hypomineralisation, such as post-eruptive breakdown, hypersensitivity, changes in enamel texture and hardness, and abnormal translucency on radiographs.
* The affected tooth is classified as having moderate or severe discolouration according to Dean's fluorosis index (Dean, 1942)
* The affected tooth has lost less than one-third of its coronal crown structure
* The affected tooth has a fracture located at the subgingival margin
* The affected tooth requires splinting due to the severity of the trauma
* Presence of severe malocclusion that could compromise the integrity of the restoration

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged 6-15 years who visit the Pediatric Dental Clinic at the Faculty of Dentistry, Mahidol University, for maxillary anterior tooth restoration
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Colour matching | Immediate, 1-week, 6-month, 12-month after restoration
  Colour match and translucency grading of 'very good' according to FDI criteria indicates clinically excellent colour matching and translucency.
Colour stability | 1-week, 6-month, 12-month after restoration
  Colour match and translucency, surface and margin staining, and surface lustre grading of 'very good' according to FDI criteria indicates clinically excellent colour stability.

SECONDARY OUTCOMES:
Patient satisfaction | 1-week, 6-month, 12-month after restoration
  Patients show the highest aesthetic satisfaction if they score 5 on a 5-point Likert scale on the aesthetic questionnaire, ranging from 5 (most satisfied) to 1 (not satisfied).
Parent satisfaction | 1-week, 6-month, 12-month after restoration
  Parents show the highest aesthetic satisfaction if they score 5 on a 5-point Likert scale on the aesthetic questionnaire, ranging from 5 (most satisfied) to 1 (not satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Pipop Saikaew, PhD, Study Director — Department of Operative Dentistry and Endodontics, Faculty of Dentistry, Mahidol University
Locations (1):
- Pediatric Dental Clinic, Faculty of Dentistry, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No